CLINICAL TRIAL: NCT04047615
Title: The Effects of an Exercise Intervention Programme on Behaviour and Fitness Levels in Children With ASD.
Brief Title: The Effects of Exercise on Behavior and Fitness in Children With ASD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institute of Technology, Carlow (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASD Intervention
Record Dates: First submitted 2019-08-05; First posted 2019-08-07 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Autism Spectrum Disorder; Behavior
MeSH Terms: conditions — Autism Spectrum Disorder; Behavior | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise effects on Behavior (Experimental): An exercise intervention programme will be implemented 3 times a week for an 8 week period of time in a school setting. Each exercise class will last 60 minutes. The exercise classes will be fun for the students to participate in and will involve aspects of fundamental movement skills.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — An exercise intervention programme will be delivered in each school for an 8 week period. Exercise classes will take place 3 times a week and will be of 60 minutes duration.

SUMMARY:
This study will examine the effects of a school based exercise intervention programme on the behaviour and fitness levels in children with autism.

DETAILED DESCRIPTION:
This study will examine the effects of a school based exercise intervention programme on the behaviour and fitness levels in children with autism. Local primary schools who have an Autism Spectrum Disorder (ASD) class will be approached to participate in the project. The age profile of the children will be 4-12 years of age and they will have mild-sever levels of autism. The exercise intervention programme will be delivered 3 times per week in the schools over an 8 week period.

Children will be fitness tested to assess the change in fitness levels over the 8 week period. Questionnaires will be given to the parents and teachers of the children at the beginning and at the end of the programme to assess changes in behaviour levels as a result of the exercise intervention programme.

ELIGIBILITY:
Inclusion Criteria:

• Diagnosis of Autism Spectrum Disorder

Exclusion Criteria:

• Any medical condition which excludes the child from partaking in exercise

Ages: 4 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2021-02 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Behavior | Change from baseline at Week 4 and Week 8
  Changes in behavior levels of the children will be assessed using the Aberrant Behavior Checklist and
Behavior | Change from baseline at Week 4 and Week 8
  Changes in behavior levels of the children will be assessed using the Gilliam Autism Rating Scale 2nd Edition.
  Higher the value (total score) the more likely the individual has Autism.

SECONDARY OUTCOMES:
Fitness Level | Change from baseline at Wkke 4 and Week 8
  The modified eurofit test will be used to investigate fitness levels of the children

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Technology, Carlow, Carlow, Ireland